CLINICAL TRIAL: NCT01199744
Title: Collection of Patients' Background InformationRelenza® Sentinel Site Monitoring Program in Japan
Brief Title: Relenza® Sentinel Site Monitoring Program in Japan
Acronym: SSMP
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114045
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Influenza, Human
Keywords: Influenza; Relenza®; SSMP
MeSH Terms: conditions — Influenza, Human | interventions — Zanamivir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Influenza virus infection patients exposed to zanamivir: Safety of Influenza virus infection patients exposed to zanamivir
  Interventions: Drug: zanamivir

INTERVENTIONS:
Drug: zanamivir — zanamivir

SUMMARY:
To collect background information of patients receiving a prescription for Relenza® and study risk factors etc. for adverse drug reactions collected through spontaneous reporting. In particular, to characterize the types and incidences of adverse events, serious adverse events, and adverse drug reactions and to investigate risk factors for them in patient populations that are regarded to be at high risk for novel influenza A (H1N1)and in which the use experience of Relenza® has not been enough (such as pregnant women, infants, elderly persons, and those with decreased physical function) in accordance with the PFSB/SD Notification 0904, No.2 of the Safety Division, Pharmaceutical and Food Safety Bureau, MHLW, dated 4th September 2009.

To compare the data with the safety data collected in overseas sentinel site monitoring programs.

DETAILED DESCRIPTION:
1. Objectives To collect background information of patients receiving a prescription for Relenza® and study risk factors etc. for adverse drug reactions collected through spontaneous reporting. In particular, to characterize the types and incidences of adverse events, serious adverse events, and adverse drug reactions and to investigate risk factors for them in patient populations that are regarded to be at high risk for novel influenza A (H1N1)and in which the use experience of Relenza® has not been enough (such as pregnant women, infants, elderly persons, and those with decreased physical function) in accordance with the PFSB/SD Notification 0904, No.2 of the Safety Division, Pharmaceutical and Food Safety Bureau, MHLW, dated 4th September 2009.

   To compare the data with the safety data collected in overseas sentinel site monitoring programs.
2. Planned number of patients Planned number of patients: 1,600 cases (of which 90 shall be pregnant women)
3. Target patients All patients who visit a sentinel site between the date of the contract and 31st March 2010 and are prescribed Relenza® for the purpose of either treatment or prophylaxis of influenza.
4. Planned number of sentinel sites About 20 sites, mainly obstetrics, pediatrics, and internal medicine.
5. Method 1)The sentinel sites to participate in the monitoring program will be selected from medical institutions which has adopted/purchased Relenza®. Physicians who are capable of fulfilling the objectives of the program satisfactorily will be given information concerning the purpose, target patients, data to be collected, method, etc. and asked for cooperation.

2)Upon receiving consent of the physician for cooperation, a written contract will be concluded with the head of the site (e.g., hospital director) before collection of patient background information is started.

3)All patients receiving a prescription of Relenza® during the contract term at the respective site (i.e., from the date of contract until 31st March 2010) will be included in the monitoring program. At sentinel sites with obstetrics service, all pregnant women receiving a prescription of Relenza® during the contract term at the respective site (i.e., from the date of contract until 31st March 2010) will be included in the monitoring program in order to focus on collection of data in pregnant women.

4)Physician in charge will enter the data such as the background information of the patients who have received prescription of Relenza® from the date of contract until 31st March 2010 into the electronic data collection (EDC) system, check the data, and transmit them to GlaxoSmithKline K.K.

5)The period of observation is 11 days after prescription of Relenza®. 6)Information about cases with adverse events and use of Relenza® during pregnancy shall be reported separately through spontaneous ADR reporting system.

6.Planned monitoring period November 2009 to 31st March 2010 The data collection will be concluded before 31st March 2010 when the requisite number of patients is accrued ahead of schedule.

7.Data to be collected

1. Patient identification number to identify each patient.
2. Reason for the use of Relenza® (prophylaxis or treatment); if Relenza® is used for the treatment: information whether or not influenza virus test was performed in the clinical laboratory; if yes, result of the influenza virus test (Pandemic Flu (H1N1) or Seasonal Flu).
3. Patient background information : Birth year, sex (if female: pregnant or not pregnant, breastfeeding or not breastfeeding), body height, body weight, complications (if yes: bronchial asthma, chronic obstructive pulmonary disease, immune deficiency disease [if yes: HIV infection, organ transplant, congenital immunodeficiency, hematological malignancy, autoimmune disease, chemotherapy], others), route of infection (family infection or group infection), influenza vaccination status (if vaccinated: date of vaccination, generic name or brand name of the vaccine used).
4. Prescription information for Relenza®: Relenza® dose, dosing frequency per day, Relenza® initiation date, last date of administration)
5. Date of patient contact; was a contact with the patient established? (if yes, type of contact [telephone, e-mail, in person]).
6. Adverse events information If adverse events are reported, information concerning the circumstance of the adverse event shall be reported separately in the form of spontaneous reporting.
7. Concomitant medications during Relenza® treatment (generic name or trade name of the drug, reason for the use of the drug, dose, dosing frequency per day, unit, initiation date, last date of administration, still on the medication, use for the treatment of adverse event)
8. Completion or discontinuation of data collection
9. If Relenza® is used during pregnancy, the course of pregnancy and delivery, abortion, etc. adverse events observed in mother and/or infant shall be reported separa

ELIGIBILITY:
Inclusion Criteria:

Prescribed Relenza® for the purpose of either treatment or prophylaxis of influenza

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1600 cases (of which 90 shall be pregnant women)
Sampling Method: Probability Sample
Enrollment: 1575 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Medicine and Drug Journal Vol.46 No.12 p.136-142, 2010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Sentinel Site Monitoring Program collected the patient background and safety data of Relenza administered in the Japanese population per the requirements of the Japanese Ministry of Health, Labour and Welfare (MHLW).
Groups:
- Relenza: Dose and frequency of dosing was based on prescribing information. Treatment dose: 10 milligrams (mg) twice daily for 10 days. Prophylactic dose: 10 mg once daily for 10 days.
Period: Overall Study
Arm/Group | Relenza
Started | 1575
Completed | 1575
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Relenza
Number analyzed (Participants) | 1575
Age, Customized [Number; unit: participants]
  >=3 to <7 years | 195
  >=7 to <15 years | 790
  >=15 to <65 years | 586
  >=65 to <74 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 827
  Male | 748

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Drug Reaction
Description: An adverse drug reaction is defined as a drug adverse event that a physician has determined to be related to the use of Relenza. A drug adverse event is defined as any unfavorable or unintended sign (including laboratory test abnormalities), symptom, or disease that occurs when a drug is administered, regardless of the relationship to the drug. For a complete list of all adverse drug reactions recorded during the study, see the section entitled "Other (Non-serious) Adverse Events."
Time Frame: 5 months (November 2009 to March 2010)
Population: All participants who visited the sentinel 26 centers from the date of the contract to 31st March 2010 and were prescribed Relenza for the purpose of either treatment or prophylaxis of influenza
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants | 4

2. Secondary Outcome: Number of Participants With Any Serious Adverse Drug Reaction (ADR)
Description: A serious ADR is defined as a serious adverse drug event (ADE) that a physician has determined to be related to the use of Relenza. Serious ADE: death caused by an ADR; an event that is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in severe symptoms requiring treatment so that symptoms do not lead to previously mentioned outcomes, and a congenital anomaly/birth defect. For a complete list of all serious ADRs recorded during the study, see "Serious Adverse Events" section.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants | 1

3. Secondary Outcome: Number of Male and Female Participants With Either a Serious or Non-serious Adverse Drug Reaction
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Male | 3
  Female | 1

4. Secondary Outcome: Number of Participants in the Indicated Age Categories With Either a Serious or Non-serious Adverse Drug Reaction
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  >=3 to <7 years | 0
  >=7 to <15 years | 3
  >=15 to <65 years | 1
  >=65 to <74 years | 0

5. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Categorized by Reason for the Use of Relenza
Description: The dose given for treatment of influenza is 10 mg twice daily for 5days. Prophylaxis is defined as a measure taken for the prevention of a disease or condition. The prophylactic dose of Relenza is 10 mg once daily for 10 days.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Treatment | 4
  Prophylaxis | 0

6. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Categorized by Either Having Complications or Having no Complications
Description: A complication is defined as asthma.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Complications | 1
  No complications | 3

7. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Categorized by Either Having Risk Factors for Influenza or Having no Risk Factors
Description: Risk factors are defined as pregnancy; infancy; being elderly; and having chronic respiratory disease, cardiocirculatory disease, and/or diabetes.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Risk factor | 1
  No risk factor | 3

8. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Who Were Also in the Indicated High-risk Categories
Description: Participants with only hypertension were excluded from the cardiocirculatory disease category. Participants in high-risk categories are at risk for the aggravation of both infection and symptoms.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Pregnant | 0
  Infant (<7 years of age) | 0
  Elderly (>=65 years of age) | 0
  Chronic respiratory disease | 1
  Cardiocirculatory disease | 0
  Diabetes | 0

9. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Who Were Vaccinated for Influenza
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Vaccinated | 1
  Not vaccinated | 3

10. Secondary Outcome: Number of Participants With Either a Serious or Non-serious Adverse Drug Reaction Who Were Also Taking Concomitant Medications
Description: Concomitant medications are defined as drugs used during the administration of Relenza.
Time Frame: 5 months (November 2009 to March 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Relenza
Number analyzed (Participants) | 1575
participants
  Concomitant medication | 4
  No concomitant medication | 0

ADVERSE EVENTS:
Arm/Group | Relenza
Serious Adverse Events (participants affected / at risk) | 1/1575
Other Adverse Events (participants affected / at risk) | 4/1575
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relenza (N=1575)
Depressed level of consciousness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relenza (N=1575)
Abnormal behavior (Psychiatric disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.